CLINICAL TRIAL: NCT05530590
Title: Training the Long-Term Services and Supports Dementia Care Workforce in Provision of Care to Sexual and Gender Minority Residents
Brief Title: Minnesota Inclusive LTSS for LGBTQ Seniors
Acronym: MILLS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00014177; 5R01AG075734 (NIH)
Record Dates: First submitted 2022-07-22; First posted 2022-09-07 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Long-term support and service facilities; Alzheimer Disease; Dementia; LTSS; Seniors
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: The study involves conducting a 3-arm, stratified (management/staff), group (agency) randomized controlled trial (RCT) of the in-person vs. online intervention vs. waitlist control on organizational factors (i.e., environment and policy) and on staff knowledge, attitudes, and skills.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training to Serve (TTS) in person training (Experimental): Participants are provided access to the pretest one week before the training. On the day of training, when the trainers arrive, participants have a final opportunity to complete the baseline survey before the intervention. Tablets will be available to complete pre- and post- surveys. The training for management takes 3-4 hours, and for staff, one hour. For consistency and feasibility, both trainings are conducted by the same trainers at the same visit. Immediately after the intervention, participants complete the post-intervention seminar evaluation assessing knowledge and attitudes/comfort in serving SGM clients.
  Interventions: Other: Training to Serve (TTS) in person training
- Training to Serve online training (eTTS) (Experimental): Participants are provided a unique identifier to access the online website. The opening page welcomes them to the study, then directs them to the chunked consent materials and baseline survey. As soon as they have completed this, they receive access to the intervention, which for management is expected to take 1-2 hours and for staff, 30-45 minutes (i.e., the online equivalent of 3-4 and 1 hour, respectively). After completion of the required modules, participants receive access to the optional modules as well as the posttest survey to evaluate the training. Once the post-test is complete, they are thanked for their involvement and informed they will receive an e-mail to access a follow-up survey in six months' time.
  Interventions: Other: Training to Serve online training (eTTS)
- Waitlist control (No Intervention): Participants complete the baseline survey, then they receive a note thanking them for completing all activities and informing them the intervention will be available in 6 months' time.

INTERVENTIONS:
Other: Training to Serve (TTS) in person training — Participants receive in person training.
  Arms: Training to Serve (TTS) in person training
Other: Training to Serve online training (eTTS) — Participants receive online training.
  Arms: Training to Serve online training (eTTS)

SUMMARY:
This study is designed to help improve the care of sexual and gender minority (SGM) with Alzheimer's Disease and Alzheimer's Disease Related Dementia (AD/ADRD) in long-term services and supports (LTSS) by training the state's LTSS workforce in SGM culturally responsive care. The randomized controlled trial will rigorously test the effects of an in person versus an online training program on improving SGM culturally responsive care with a waitlist control.

DETAILED DESCRIPTION:
The study involves conducting a 3-arm, stratified (management/staff), group (agency) randomized controlled trial (RCT) of the in-person vs. online intervention vs. waitlist control on organizational factors (i.e., environment and policy) and on staff knowledge, attitudes, and skills.

ELIGIBILITY:
Inclusion Criteria:

* licensure in Minnesota to provide nursing and/or as a housing with services establishment
* Willingness to undertake a policy and environment review at baseline and 6 months later
* having at least 5 managers/ supervisors and 5 staff.

Exclusion Criteria:

* Participants who cannot speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-04-21 (Estimated); Study Completion 2026-07-04 (Estimated)

PRIMARY OUTCOMES:
Environment change | baseline and 6-months follow up
  Access to sexual and gender minority (SGM) providers, gender neutral intake forms
Skills assessment | Baseline
  Ability to conduct 7 skills key to providing competent care to SGM
Skills assessment | Immediately post-intervention
  Ability to conduct 7 skills key to providing competent care to SGM
Competence in SGM Care | 6 months after intervention
  Competent scale when it comes to providing care to SGM

SECONDARY OUTCOMES:
SGM with AD/ADRD referenced explicitly in policies | Baseline
  Human Resources policies and intake forms
SGM with AD/ADRD referenced explicitly in policies | 6 months post-intervention
  HR policies and intake forms
SGM knowledge | Baseline
  10-item review of key content in training
SGM knowledge | immediately post-intervention
  10-item review of key content in training
SGM knowledge | 6 months post-intervention
  10-item review of key content in training
SGM attitudes | Baseline
  Homonegativity scale
SGM attitudes | immediately post-intervention
  Homonegativity scale
SGM attitudes | 6 months post-intervention
  Homonegativity scale
Health care empathy | Baseline
  Jefferson Physician Empathy student version
Health care empathy | immediately post-intervention
  Jefferson Physician Empathy student version
Health care empathy | 6 months post-intervention
  Jefferson Physician Empathy student version

OTHER OUTCOMES:
Discrimination experience at work | Baseline
  Adapted everyday discrimination scale
Discrimination experience at work | immediately post-intervention
  Adapted everyday discrimination scale
Discrimination experience at work | 6 months post-intervention
  Adapted everyday discrimination scale
Social desirability at work | Baseline
  Marlowe Crowne Social desirability scale
Social desirability at work | immediately post-intervention
  Marlowe Crowne Social desirability scale
Social desirability at work | 6 months post-intervention
  Marlowe Crowne Social desirability scale
Sexual and Religious Identification | Baseline
  Duke Religiosity Index
Sexual and Religious Identification | 6 months follow-up post-intervention
  Duke Religiosity Index
Agency demographics | Baseline
  Agency type, size and staff
SGM estimate | Baseline and 6 month follow up.
  Number of SGM staff
SGM estimate | 6 months follow up post-intervention
  Number of SGM staff

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rosser, PhD,MPH, Principal Investigator — University of Minnesota; Tetyanna Shippee, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No